CLINICAL TRIAL: NCT02202681
Title: Pilot Study for Imaging of the Duodenum Using an OFDI Capsule
Brief Title: Imaging the Duodenum Using an Optical Frequency Domain Imaging OFDI Capsule
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-P001405
Record Dates: First submitted 2014-06-12; First posted 2014-07-29 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Celiac Disease; Healthy
Keywords: Duodenum; Optical Frequency Domain Imaging (OFDI); Optical Coherence Tomography; Imaging; Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OFDI Capsule Imaging (Experimental): Participant will swallow the OFDI Capsule and imaging will be performed using the OFDI system.
  Interventions: Device: OFDI Capsule

INTERVENTIONS:
Device: OFDI Capsule — Imaging of the duodenum with the OFDI capsule and system

SUMMARY:
The study is being done to assess the tolerability and feasibility of a tethered OFDI capsule to image the duodenum.

A total of 108 participants (36 healthy and 72 with clinically suspected or diagnosed Celiac disease) will be asked to swallow the tethered capsule, while they are awake and unsedated and ask for their feedback. Images will be taken using the OFDI system while the capsule travels from the esophagus into the stomach and into the duodenum.

DETAILED DESCRIPTION:
Participants including healthy volunteers as well as patients with Celiac disease will be recruited and asked to swallow the OFDI capsule while being awake and unsedated. The capsule is attached to a tether which allows the operator to control as well as navigate the capsule as it progresses down the esophagus, through the stomach and into the duodenum using natural propulsive force called peristalsis.

As the capsule progresses, multiple 2-dimensional cross-sectional images of the duodenum are acquired. Images are analyzed at a later stage.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be over 18 years for healthy volunteers
* Participants must be over 16 years for patients with Celiac disease
* Participant must be able to give informed consent

Exclusion Criteria:

* Participants with an inability to swallow pills or capsules.
* Participants with esophageal or intestinal fistulas.
* Participants with known esophageal or intestinal strictures resulting in a luminal diameter smaller than the diameter of the capsule.
* Participants with a history of intestinal Crohn's disease.
* Women who are pregnant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2013-09-16 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Tolerability of OFDI Imaging in subjects swallowing the OFDI capsule | Images will be acquired during the OFDI imaging session which should on average take anywhere from 30 minutes to 2 hours.
  After participating in the study, the participant will be asked for feedback about tolerability of the procedure using a questionnaire.
Feasibility of OFDI Imaging in subjects swallowing the OFDI capsule | Images will be acquired during the OFDI imaging session which should on average take anywhere from 30 minutes to 2 hours
  An investigator will assess the quality of the recorded images and movies obtained with each exam after the imaging is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No